CLINICAL TRIAL: NCT07004647
Title: An Investigator-Initiated, Single-Arm, Dose-Escalation Exploratory Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Preliminary Efficacy of MT027 Cell Injection in Patients With Advanced Primary or Secondary Peritoneal Tumors
Brief Title: MT027 Cell Injection in Patients With Advanced Primary or Secondary Peritoneal Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT027-PNT-003
Record Dates: First submitted 2025-04-14; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Peritoneal Tumor
MeSH Terms: interventions — fludarabine

STUDY DESIGN:
Intervention Model Description: Accelerated titration and 3+3 design dose escalation phase followed by dose expansion phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MT027 Cell injection (Targeting B7-H3 Generic generic chimeric antigen receptor T cell injection). (Experimental)
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — D-10 to D-2: Fludarabine (25 mg/m2/day) will be administered intravenously for 3 days;D-10 to D-2: Cyclophosphamide (250 mg/m2/day) will be administered intravenously for 3 days.

SUMMARY:
This study is a single-arm, dose-escalation, investigator-initiated exploratory clinical trial designed to evaluate the tolerability, safety, pharmacokinetic profile, and preliminary efficacy of MT027 Cell Injection in patients with advanced primary or secondary peritoneal tumors.

DETAILED DESCRIPTION:
This study evaluates the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of intrathecal or intracerebroventricular (ICV) injection of MT027 in glioma treatment. Partial clinical data have been presented at the 2024 ASCO Annual Meeting. Dose Groups: Three predefined dose levels: 1×10⁷ cells/dose、3×10⁷ cells/dose、6×10⁷ cells/dose. Administration frequency: Every 2 weeks (with a 4-week dose-limiting toxicity [DLT] observation period after the first injection, followed by subsequent injections every 2 weeks). Dose Escalation: Accelerated titration + 3+3 design: First dose cohort: Accelerated titration strategy. Subsequent cohorts: Standard "3+3" dose-escalation. Dose Adjustment: After reaching predefined dose levels, if no DLT or significant safety events occur, dose escalation decisions (including MTD determination) will be jointly reviewed by investigators and collaborators based on integrated safety and efficacy data. Primary Objectives: To assess the safety, tolerability, and determine the maximum tolerated dose (MTD) of MT027 cell injection in patients with advanced primary or secondary peritoneal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in this study and provision of a signed and dated written informed consent form before any study-specific procedures, sampling or analysis are conducted;
* Age range: 18 to 70 years old (inclusive), gender unrestricted
* Confirmed diagnosis of primary peritoneal tumors (including primary peritoneal carcinoma and malignant peritoneal mesothelioma) by cytological and/or histological methods, supported by complete pathological report documentation, with failure of first-line standard therapy.
* Patients with secondary peritoneal tumors confirmed by cytological and/or histological diagnosis (e.g., secondary to adenocarcinomas of gastric, colorectal, platinum-resistant advanced ovarian, or fallopian tube origin) who meet the following criteria: Treatment Failure: Progression after ≥2 prior lines of standard therapy; Lack of Standard Options: No available standard treatment, and/or Intolerance to Standard Therapy: Defined as: Grade ≥3 adverse events (AEs) related to prior therapy, or Persistent/recurrent AEs below grade 3 that preclude further treatment (as judged by the investigator).

  *：Patients with pseudomyxoma peritonei (PMP) of ovarian or appendiceal origin will be excluded from this study.
* Contrast-enhanced CT/MRI demonstrating intra-abdominal space-occupying lesions with at least one evaluable target lesion (per iRECIST criteria);
* Prior to enrollment, systemic anti-tumor therapies must meet the following washout period requirements:

  1. Nitrosoureas and mitomycin C: ≥6 weeks;
  2. Other chemotherapeutic agents and small-molecule targeted agents: ≥3 weeks or • half-lives (including active metabolites), whichever is longer;
  3. Biological agents (such as immune checkpoint suppression), ≥4 weeks;
  4. Biologics (e.g., immune checkpoint inhibitors): ≥4 weeks
* Subjects must meet **one** of the following criteria: Willing to provide either: FFPE tissue blocks or 8 consecutive unstained slides from the most recent pathological specimen, or Ascites tumor cells (for cytological analysis), with B7-H3 positivity confirmed in the tumor tissue/ascites; OR Documented B7-H3 positivity in archival tumor tissue (e.g., from prior immunohistochemistry or RNA-seq reports).
* No intraperitoneal drug injections (including hyperthermic intraperitoneal chemotherapy, HIPEC) have been administered within 1 month prior to signing the informed consent form, except for diagnostic paracentesis.;
* Life expectancy ≥3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-2;
* Laboratory tests during the screening period must meet the following criteria (no blood transfusion, G-CSF use, or medication to correct values within 14 days prior to hematological testing) :
* Blood routine (within 7 days) :
* White Blood Cells (WBC) ≥3.0×10⁹/L;
* Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L;
* Lymphocytes ≥0.8×10⁹/L;
* Platelets (PLT) ≥90×10⁹/L;
* Hemoglobin (HGB)≥90 g/L (*transfusion and erythropoietin use are permitted*); If active bleeding or other ongoing conditions (e.g., hemolysis, bone marrow infiltration) lead to increased red blood cell destruction/impaired production, requiring repeated transfusions or erythrocyte therapies, the patient's eligibility must be discussed with the **sponsor** based on clinical context prior to enrollment.
* Liver function (within 7 days) :
* Total Bilirubin (TBIL) ≤1.5× upper limit of normal (ULN);
* ALT/AST≤2.5× ULN;
* Kidney function (within 7 days) :
* Serum Creatinine (Cr)≤1.5× ULN or Creatinine Clearance (CrCl) ≥30 mL/min (calculated by Cockcroft-Gault formula) Cockcroft-Gault formula);
* Coagulation function (within 7 days) :
* International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5× ULN;
* Activated Partial Thromboplastin Time (APTT) ≤1.5× ULN;
* Toxicities from prior systemic therapy must have recovered to≤ Grade 1 or baseline levels prior to the first dose (except for alopecia);
* Males of reproductive potential and females of childbearing potential must agree to use highly effective contraception from the time of signing the informed consent form until 180 days after the last dose of MT027 Cell Infusion. Females of childbearing potential include: Premenopausal women .Women within 2 years postmenopausal.

Exclusion Criteria:

* Known hypersensitivity to the investigational product or its excipients;
* Other malignancies within 5 years (except cured carcinoma in situ of cervix/breast/prostate/thyroid/skin [basal cell/squamous cell carcinoma]);
* Contraindications to peritoneal puncture or investigator-determined unsuitability for intraperitoneal therapy;
* MSI-H (microsatellite instability-high)/dMMR (mismatch repair deficient) colorectal cancer patients without prior immunotherapy;
* Portal vein thrombosis confirmed by imaging;
* Bowel obstruction within 4 weeks prior to dosing;
* Peritoneal adhesions/jelly-like ascites (e.g., pseudomyxoma peritonei) limiting drug diffusion;
* Major surgery (except intraperitoneal port placement) or abdominal radiotherapy within 4 weeks before first dose;
* High-dose systemic corticosteroids (prednisone ≥20 mg/day) for >14 days within 4 weeks prior to treatment (topical/inhaled steroids allowed);
* Participation in other clinical trials within 4 weeks prior to screening;
* Prior therapy targeting same pathway (antibody/ADC/cell therapy);
* Severe autoimmune diseases (e.g., lupus, rheumatoid arthritis);
* Recipients of allogeneic tissue/organ transplants;
* Live vaccination within 4 weeks before cell therapy or planned during study;
* Active infections: HBV (HBsAg+ with detectable DNA)、 HCV (Ab+ except RNA-undetectable) 、 HIV+ 、Syphilis (TPPA+) 、Active EBV/CMV infection;
* Active systemic infections, coagulopathy, or other significant comorbidities;
* Organ dysfunction: Cardiac: NYHA Class ≥III ；Hepatic: Child-Pugh C； Renal: CKD Stage ≥4 ；Pulmonary: Severe respiratory failure;
* Pregnancy/Lactation;
* Investigator-determined unsuitability based on clinical/laboratory findings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 2 years
  Incidence and severity of adverse events.
Serious Adverse Events (SAEs) | 2 years
  Incidence and severity of serious adverse events.
Adverse Events of Special Interest (AESI) | 2 years
  Adverse Events of Special Interest (AESI)(Incidence and severity ) Incidence and severity of adverse event of special interest.
Identification of Maximum Tolerated Dose (MTD) & Incidence of Dose-limiting Toxicities (DLTs) | 4 weeks after the CAR-T cells infusion
  Incidence and severity of dose-limiting toxicities (DLTs) following infusion of CAR-T cell injection, at each dose level tested in dose escalation phase.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The Objective Response Rate (ORR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Disease Control Rate (DCR) | 2 years
  Disease control rate (DCR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.
Duration of Overall Response (DOR) | 2 years
  Time from documentation of disease response to disease progression.
Progression-Free Survival (PFS) | 2 years
  PFS is defined as the time from CAR-T infusion to the date of the disease progression or death from any cause.
Overall Survival (OS) | 2 years
  OS is defined as the time from CAR-T infusion to the date of death due to any cause.
Bio-distribution of Anti mesothelin CAR-T cells | 2 years
  CAR copies will be measured by qPCR to evaluate the expansion and persistenc e of CAR-T cells in vivo. Cmax, Tmax, AUC0-tlast and AUC0-inf of CAR copies will be analyzed.
  Cmax is the maximum CAR level in peripheral blood or bone marrow. Tmax is time to peak CAR level in blood or bone marrow. AUC0-tlast and AUC0-inf are area under the curve of the CAR level in blood .
Cytokine Level in Peripheral Blood | 2 years
  Level of cytokines in serum.
Anti-drug Antibodies | 2 years
  Number of participants with anti-drug antibodies.
RP2D | 4 weeks after the CAR-T cells infusion
  The RP2D is the optimal dose level selected for further evaluation in Phase II clinical trials, based on safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and preliminary efficacy data gathered during Phase I dose-escalation studies. It represents the dose that balances maximum therapeutic benefit with acceptable toxicity for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China